CLINICAL TRIAL: NCT05165940
Title: Improving Care for Veterans by Understanding and Facilitating Transition to Recommended PTSD Treatment (CDA 21-194)
Brief Title: Facilitating Transition to Recommended PTSD Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CDX 22-002; 1IK2HX003339-01A2 (NIH)
Record Dates: First submitted 2021-12-02; First posted 2021-12-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: PTSD
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive care coordination as usual (i.e., TAU) through the VA or an experimental care coordination intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAU (Active Comparator): Treatment As Usual with a VA mental health treatment coordinator
  Interventions: Behavioral: Treatment As Usual
- New Health Services Intervention (Experimental): Novel health services intervention with a VA mental health treatment coordinator
  Interventions: Behavioral: New Health Services Intervention

INTERVENTIONS:
Behavioral: Treatment As Usual — Care Coordination Treatment as usual with a VA mental health treatment coordinator
  Arms: TAU
Behavioral: New Health Services Intervention — The experimental care coordination intervention begins with a 60-minute in-person session and continues with regular, brief contacts between the Veteran and clinician. During the first session, the clinician and Veteran will (1) discuss the Veteran's beliefs about their presenting problem; (2) collaboratively identify SMART goals; (3) discuss treatment options; (4) use shared decision-making to match treatment to SMART goals; (5) develop criteria to evaluate treatment progress; and (6) manage treatment expectations. During follow-up sessions, the clinician and Veteran will reflect on treatment progress, make appropriate updates to SMART goals, and re-evaluate barriers to CPT or PE.
  Arms: New Health Services Intervention

SUMMARY:
Cognitive processing therapy (CPT) and prolonged exposure therapy (PE) were widely disseminated as recommended posttraumatic stress disorder (PTSD) treatments. However, post-9/11 Veterans with PTSD rarely initiate CPT or PE, especially as an initial treatment. Little research has explored the combinations and sequences of psychosocial and medication treatments that Veterans receive ("treatment sequences"). One common and understudied treatment sequence begins with stabilization treatment, which is designed to prepare Veterans for CPT or PE. There is a significant research gap in understanding how treatment sequence affects initiation of CPT or PE. The proposed research is an innovative, mixed-methods approach to assessing the impact of variability in treatment sequence, including stabilization treatment, on initiation of CPT or PE and applying this knowledge by developing a health services intervention that facilitates timely transition to CPT or PE. Research aims can improve PTSD treatment by increasing initiation of and reducing disparities in CPT/PE.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is one of the most common mental health diagnoses among Veterans. Cognitive processing therapy (CPT) and prolonged exposure therapy (PE) were widely disseminated in the Veterans Health Administration (VHA) as recommended PTSD treatments. Despite these efforts, few post-9/11 Veterans diagnosed with PTSD initiate CPT or PE. In the small percentage of Veterans who receive these therapies, CPT and PE are rarely the first treatment a Veteran receives. A common treatment sequence identified in implementation research, begins with "stabilization treatment," combinations of psychosocial and medication treatments that prepare Veterans for CPT or PE. Despite consistently identifying stabilization treatment as a common VHA practice, little research has investigated this treatment sequence. A novel approach to solving existing limitations in PTSD treatment delivery involves developing an intervention that both acknowledges the ubiquitous presence and benefits of stabilization treatment, while facilitating timely transition from stabilization treatment to CPT or PE. This CDA-2 aims to improve delivery of PTSD services in the VHA. The proposed research aims are: (1) To qualitatively understand Veterans' and clinicians' perspectives on selecting stabilization treatments and how stabilization treatment serves as a barrier or facilitator of transition to CPT or PE; (2) To develop and conduct a randomized, pragmatic pilot trial of a brief, Veteran-centered intervention to support transition from stabilization treatment to CPT or PE; and (3) To identify sociodemographic disparities in treatment sequences and to determine how treatment sequences influence time to CPT or PE initiation across the VHA.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Diagnosed with PTSD as part of an intake assessment at the San Francisco Veterans Affairs Medical Center.

Exclusion Criteria:

* Inability to provide informed consent
* Cognitive impairment that precludes comprehension of study materials
* Active psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-05-03 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Initiation of Recommended PTSD Treatment | Through study completion, an average of 1 year
  Patient self-report or documentation in the electronic health record of initiating either cognitive processing therapy (CPT) or prolonged exposure therapy (PE).

SECONDARY OUTCOMES:
Acceptability (Discontinuation of Mental Health Treatment without Provider Concurrence) | Through study completion, an average of 1 year
  Patient self-report or documentation in the electronic health record that a patient has discontinued all mental health treatment without provider concurrence.
Limited Efficacy Testing (PTSD Symptom Severity) | Through study completion, an average of 1 year
  Self-Reported PTSD Symptom Severity as assessed by the PTSD Checklist for DSM-5.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Holder, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No